CLINICAL TRIAL: NCT04741334
Title: Mild Head Injury and Oral Anticoagulants: a Prospective Observational Study
Brief Title: Mild Head Injury, Antiplatelets, and Anticoagulants
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CANDELLI MARCELLO, Adjunct Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 36042/19 2721
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Craniocerebral Trauma; Cerebral Hemorrhage
Keywords: Mild head injury; Traumatic cerebral hemorrhage; Direct anticoagulants drugs; Antiplatelets drugs
MeSH Terms: conditions — Craniocerebral Trauma; Cerebral Hemorrhage; Cerebral Hemorrhage, Traumatic | interventions — Factor Xa Inhibitors; Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients not in therapy with anticoagulants or antiplatelets drugs: Patients presenting in ED with mild head trauma and not in therapy with antiplatelets and/or anticoagulants
- patients in therapy with direct anticoagulant: Patients presenting in ED with mild head trauma and in therapy with direct anticoagulants
  Interventions: Drug: direct anticoagulant
- patients in therapy with oral anticoagulant (dicumarolics): Patients presenting in ED with mild head trauma and in therapy with oral anticoagulants (dicumarols)
  Interventions: Drug: Dicumarols
- patients in therapy with antiplatelet drugs: Patients presenting in ED with mild head trauma and in therapy with antiplatelets
  Interventions: Drug: antiplatelet drugs

INTERVENTIONS:
Drug: direct anticoagulant — exposure to direct anticoagulant
  Other Names: DOAC
  Groups: patients in therapy with direct anticoagulant
Drug: antiplatelet drugs — exposure to antiplatelet drugs
  Groups: patients in therapy with antiplatelet drugs
Drug: Dicumarols — exposure to dicumarols
  Groups: patients in therapy with oral anticoagulant (dicumarolics)

SUMMARY:
Approximately 20% of patients with mild head injury presenting to the Emergency Department (ED) is taking antiplatelet agents and 10% is taking oral anticoagulants. The aim of the study is to determine the prevalence of cerebral hemorrhage in patients presenting to the ED with an MHI. It also aims to determine whether the use of antiplatelet agents and anticoagulants may be a risk factor for the occurrence of cerebral hemorrhage and mortality. This is a prospective observational study that will include all patients who present to ED at Gemelli Hospital for an MHI for 2 years. Patients will be divided into four groups according to whether or not they are taking anticoagulants and antiplatelet drugs. Groups will be compared to evaluate the possible increased risk of complications in patients on treatment and among the different medications.

DETAILED DESCRIPTION:
Mild head injury (MHI) is one of the most common causes of emergency department (ED) admission. Approximately 20% of MHI patients admitted to PS with a mild traumatic brain injury is taking antiplatelet medications and 10% is taking oral anticoagulants. There are a few data describing the risk of adverse events in patients with MHI taking direct oral anticoagulants (DOAC), and they are of poor quality.

The aim of this study is to investigate the prevalence of cerebral hemorrhage in patients presenting to the ED with an MHI. Moreover, it will be evaluated whether the use of antiplatelet agents and anticoagulants may be a risk factor for the occurrence of cerebral hemorrhage and mortality. This is a prospective observational study that will include all patients who present to the ED at Gemelli Hospital for an MHI for 2 years. Patients will be divided into four groups according to whether or not they are taking anticoagulants and antiplatelet agents. The investigators will then determine the prevalence of cerebral hemorrhage, the need for hospitalization or neurosurgery, and mortality at different follow-up time points for each group. The investigators will compare the groups to assess the potential increased risk in patients on treatment and among drugs.

It can be hypothesized that the use of dicumarol anticoagulants and antiplatelet agents for head injury is associated with a higher risk of cerebral hemorrhage than the use of DOACs. It may be, also, hypothesize that patients taking DOACs are at a higher risk of bleeding than patients not treated with antiplatelet/anticoagulant agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with head trauma within 6 hours from the trauma w
* Age> 17 years
* Glasgow Coma Scale (GCS) > 13

Exclusion Criteria:

* Presence of serious diseases with a potentially less than one-month prognosis (patient with trauma following syncope from severe cardiovascular disease such as pulmonary embolism, myocardial infarction, ventricular arrhythmias, aortic dissection, aortic aneurysm rupture)
* Severe trauma in other body areas (identified in the Emergency department by means of CT scan of other body areas such as chest CT, abdomen CT, total body CT).
* history of congenital or acquired coagulation disorders (Haemophiliacs, patients with severe liver cirrhosis)
* Patients undergoing dual antiplatelets drugs or combination therapy of antiplatelet and anticoagulant
* Patients presenting with a GCS>13 and with focal neurologic deficits, suspected sunken fracture, or clinical signs of skull base fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will admit all patients over 18 years of age who present to the emergency department (ED) of the Fondazione Policlinico Gemelli in Rome, who refer to mild head trauma with a Glasgow Coma Scale (GCS) > 13, and who give consent to participate in the study. In all enrolled patients, the investigator will collect blood chemistry tests, especially on coagulation parameters, history of known risk factors present at the time of trauma, data on risk factors present at physical examination, data on CT scans of the head performed during the stay at ED, data on drug therapy taken, and finally data on hospitalization and surgery. Finally, data on a possible one-month follow-up visit will be collected. The follow-up visit is recommended according to the guidelines of a subgroup of these patients. The telephone number for an interview one month after the visit to ED will be collected to evaluate the clinical outcome at 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 2127 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
early Cerebral hemorrhage | 24 hours
  Number of participants with evidence of cerebral hemorrhage at head CT scan
skull fracture | 24 hours
  Number of participants with evidence of skull fracture at head CT scan
Hospital admission | 48 hours
  Number of participants with hospital admission for head trauma complication

SECONDARY OUTCOMES:
early mortality | 24 hours
  Number of participants death from all causes at 1 days
late mortality | 30 days
  Number of participants death from all causes at 30 days
late cerebral hemorrhage | 30 days
  Number of participants with evidence of cerebral hemorrhage at head CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Candelli, MD, PhD, Principal Investigator — Fondazione Policlinico Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli - IRCCS, Roma, Rm, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months after publication
Access Criteria: By request to the corresponding author